CLINICAL TRIAL: NCT00430417
Title: A Prospective Cohort Pilot Study of Bone Metabolism in Lactating and Non-lactating Postpartum Women and Healthy Non-pregnant Women
Brief Title: Bone Metabolism and Parathyroid Hormone-related Protein (PTHrP) Lactation Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mara Horwitz, Associate Professor of Medicne, University of Pittsburgh
Other Study IDs: 0610073; R01DK073039 (NIH)
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Bone Diseases, Endocrine
Keywords: Pregnancy; Lactation; Endocrine System Diseases; MusculoSkeletal System Disease; Hormone; Physiologic Properties
MeSH Terms: conditions — Bone Diseases, Endocrine; Breast Feeding; Endocrine System Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — archival blood serum and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 3 groups: Group 1: post-partum breastfeeding women
- Group 2: Group 2: post-partum bottlefeeding women
- Group 3: Group 3: normal non-pregnant controls who are age and race-matched to Group 1

SUMMARY:
The primary aim of the study is to measure bone formation in both lactating and non-lactating post-partum women and compare these to those in healthy non-pregnant controls. The secondary aim is to obtain measurements of Parathyroid Hormone-related Protein (PTHrP), markers of bone resorption, and calcium and vitamin D metabolism in these subjects. The investigators believe that lactating women will have an increase in bone resorption but no increase in bone formation when compared to non-lactating post-partum women and normal controls.

DETAILED DESCRIPTION:
Pregnancy and lactation are both states of altered maternal calcium and bone metabolism which may have a significant impact on the development of peak bone mass. While these two states are characterized by different hormonal environments, both have been associated with significant bone loss. The maternal hormonal mechanism for providing calcium to meet the needs of the developing fetus appear to differ from those that meet the needs of lactation. During pregnancy, the 30 gm of calcium required by the fetus comes predominantly from an increase in maternal intestinal calcium absorption which is mediated by 1, 25 dihydroxy vitamin D and other factors. Several studies have measured total and free 1, 25 dihydroxy vitamin D through pregnancy and find the values nearly double. Serum Parathyroid Hormone (PTH) levels fall to about 10-30% of the mean non-pregnant value in the first trimester and then increase to the mid-normal range by term, while ionized calcium remains normal throughout pregnancy. PTHrP levels gradually increase throughout pregnancy although the source (maternal, fetal, or placental) remains unclear. Most studies of bone metabolism in humans during pregnancy have measured changes in markers of bone turnover rather than bone density to avoid radiation exposure to the fetus. These studies have been confounded by several variables such as the effects of hemodilution in pregnancy, altered glomerular filtration rates (GFR), degradation, and clearance of markers by the placenta, which may cloud the results. Some of these studies report an increase in urinary markers of bone resorption from early to mid pregnancy while bone formation markers decrease and then rise before term. Importantly, no one has assessed state-of-the-art markers of bone formation such as P1NP in pregnancy or lactation.

During lactation in humans, it is estimated that 600 to 1000 ml of milk are produced a day with daily calcium loss of 200 to 400 mg. In contrast to pregnancy, a majority of this calcium comes from demineralization of the maternal skeleton, and is probably predominately mediated by PTHrP in the setting of low estrogen. PTHrP levels are significantly higher in lactating women than non-lactating controls while intact PTH is reduced by approximately 50% during the first several months of lactation. The source of the PTHrP is likely the mammary gland, as PTHrP levels are elevated 10,000 fold in milk and circulating maternal PTHrP levels are increased further with suckling. This is also supported by a mouse model in which the tissue-specific ablation of the PTHrP gene in the lactating mammary gland resulted is a decrease in bone loss during lactation. When PTHrP enters the maternal circulation, it stimulates maternal bone resorption from the skeleton and renal tubular resorption of calcium. PTHrP indirectly suppresses PTH as ionized calcium rises to upper levels of normal. 1, 25 dihydroxy vitamin D levels fall to within the normal range during lactation, although they have been reported to be higher in lactating than non-lactating postpartum women. Intestinal absorption of calcium also returns to normal during the post-partum period. Serial bone density measurement obtained during lactation show a fall of 3-10% in trabecular bone (spine, hip, femur) with a smaller 1-2% loss at cortical bone. Both losses are far greater that than that seen in early postmenopausal women, or in women receiving gonadotropin-releasing hormone (GnRH) agonist therapy. This implies that it is not only the fall in estrogen that mediates bone loss during lactation. The bone loss during lactation seems to be transient as there is rapid recovery of bone density in postpartum women with weaning and the resumption of menses.

Markers of bone resorption have been measured in urine in several prospective studies of lactation in humans where they have been reported to be elevated 2-3 fold. However, these results may be confounded by a decrease in GFR and volume contraction that may occur during lactation compared to pregnancy. Surprisingly, more reliable markers of bone resorption measured in serum (CTX and NTX) have not been measured in a controlled lactation study. Markers of bone formation as measured by osteocalcin (Oc) and bone specific alkaline phosphatase (BSAP) have generally been reported to be higher during lactation. However, these results are difficult to interpret as BSAP is not a very sensitive marker of bone formation. Recent data has emerged suggesting that Oc may measure bone resorption as well as formation. The current most accurate measure of bone formation is serum amino-terminal telopeptides of procollagen 1 (P1NP), which has not been measured in a control study of lactating women.

This is a prospective pilot cohort study of post-partum lactating women, post-partum non-lactating women, and matched healthy controls who are not currently or have not recently been pregnant. The investigators hope to estimate the measurable differences in bone formation and resorption by comparing blood and urine samples from lactating women to non-lactating postpartum women and normal controls. 100 female volunteers between the ages of 21 and 45 years will be recruited to achieve 75 evaluable subjects or 25 in each of the three groups. There are two study visits, one at 6-8 weeks and another at 12-14 weeks postpartum. Normal controls will be seen during the follicular phase of their menstrual cycle and they will be age and race matched to the post-partum women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian, Hispanic, or Asian women between the ages of 21-45.
* Group 1: Postpartum (singleton pregnancy) women who are exclusively breastfeeding, defined as 1 or fewer bottles of supplemental formula/day.
* Group 2: Postpartum (singleton pregnancy) women who are non-lactating, which is defined as bottle-feeding or having weaned their baby from breastfeeding for at least 4 weeks prior to study.
* Group 3: Controls - Healthy, non-pregnant women who are race and age-matched to the breastfeeding women in group one. They may not have been lactating or pregnant within the last year.

Exclusion Criteria:

* Subjects with cardiac, hypertensive, vascular, renal (serum creatinine of > 1.5), pulmonary, endocrine, musculoskeletal, hepatic, hematologic, or malignant or rheumatologic disease will be excluded from the study.
* Smokers and those with a history of significant alcohol or drug abuse are excluded.
* Baseline hypertension (systolic BP > 160 mm/Hg) or hypotension (systolic BP < 90 mm/Hg).
* Subjects taking any chronic medications except stable doses of thyroid hormone, prenatal, vitamin supplements, or oral contraceptives.
* Those who have received any investigational drug in past 90 days will be excluded from the study.
* Women who are currently pregnant will be excluded from the study.
* Women who became pregnant by in vitro fertilization IVF or any hormonal manipulation (i.e. fertility drugs such as clomid) are also excluded, as they may have an altered pre-pregnant hormonal state.
* All women will have a urine pregnancy test performed at each of the two study visits and must not be pregnant in order to continue in the study.
* Subjects are not allowed to donate blood between study visits.
* In order to narrow the statistical variations in the study population, African-Americans are excluded because of demonstrated differences in renal excretion of calcium and vitamin D absorption.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: New mothers who are either almost exclusively breast feeding or bottle feeding; normal controls to match those new mothers.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Measurements of amino-terminal telopeptides of procollagen 1 (P1NP), a marker of bone formation, in lactating and non-lactating postpartum women both at 6-8 and at 12-14 weeks post-partum, and to compare these values to those of normal controls | 4 months

SECONDARY OUTCOMES:
Measurements of Parathyroid Hormone-related Protein (PTHrP), markers of bone turnover, calcium and vitamin D metabolism | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mara J Horwitz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Dobnig H, Kainer F, Stepan V, Winter R, Lipp R, Schaffer M, Kahr A, Nocnik S, Patterer G, Leb G. Elevated parathyroid hormone-related peptide levels after human gestation: relationship to changes in bone and mineral metabolism. J Clin Endocrinol Metab. 1995 Dec;80(12):3699-707. doi: 10.1210/jcem.80.12.8530622.
- [Background] Gundberg CM, Looker AC, Nieman SD, Calvo MS. Patterns of osteocalcin and bone specific alkaline phosphatase by age, gender, and race or ethnicity. Bone. 2002 Dec;31(6):703-8. doi: 10.1016/s8756-3282(02)00902-x. PMID 12531565
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Hollis BW, Garcia-Ocana A, Stewart AF. Direct comparison of sustained infusion of human parathyroid hormone-related protein-(1-36) [hPTHrP-(1-36)] versus hPTH-(1-34) on serum calcium, plasma 1,25-dihydroxyvitamin D concentrations, and fractional calcium excretion in healthy human volunteers. J Clin Endocrinol Metab. 2003 Apr;88(4):1603-9. doi: 10.1210/jc.2002-020773. PMID 12679445
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Syed MA, Garcia-Ocana A, Bisello A, Hollis BW, Rosen CJ, Wysolmerski JJ, Dann P, Gundberg C, Stewart AF. Continuous PTH and PTHrP infusion causes suppression of bone formation and discordant effects on 1,25(OH)2 vitamin D. J Bone Miner Res. 2005 Oct;20(10):1792-803. doi: 10.1359/JBMR.050602. Epub 2005 Jun 6. PMID 16160737
- [Background] Kalkwarf HJ, Specker BL, Ho M. Effects of calcium supplementation on calcium homeostasis and bone turnover in lactating women. J Clin Endocrinol Metab. 1999 Feb;84(2):464-70. doi: 10.1210/jcem.84.2.5451. PMID 10022402
- [Background] Kovacs CS. Calcium and bone metabolism during pregnancy and lactation. J Mammary Gland Biol Neoplasia. 2005 Apr;10(2):105-18. doi: 10.1007/s10911-005-5394-0. PMID 16025218
- [Background] Kovacs CS, Kronenberg HM. Maternal-fetal calcium and bone metabolism during pregnancy, puerperium, and lactation. Endocr Rev. 1997 Dec;18(6):832-72. doi: 10.1210/edrv.18.6.0319. No abstract available. PMID 9408745
- [Background] Sowers M. Pregnancy and lactation as risk factors for subsequent bone loss and osteoporosis. J Bone Miner Res. 1996 Aug;11(8):1052-60. doi: 10.1002/jbmr.5650110803. No abstract available. PMID 8854240
- [Background] Sowers M, Eyre D, Hollis BW, Randolph JF, Shapiro B, Jannausch ML, Crutchfield M. Biochemical markers of bone turnover in lactating and nonlactating postpartum women. J Clin Endocrinol Metab. 1995 Jul;80(7):2210-6. doi: 10.1210/jcem.80.7.7608281.
- [Background] Sowers MF, Hollis BW, Shapiro B, Randolph J, Janney CA, Zhang D, Schork A, Crutchfield M, Stanczyk F, Russell-Aulet M. Elevated parathyroid hormone-related peptide associated with lactation and bone density loss. JAMA. 1996 Aug 21;276(7):549-54. PMID 8709404
- [Background] VanHouten JN, Dann P, Stewart AF, Watson CJ, Pollak M, Karaplis AC, Wysolmerski JJ. Mammary-specific deletion of parathyroid hormone-related protein preserves bone mass during lactation. J Clin Invest. 2003 Nov;112(9):1429-36. doi: 10.1172/JCI19504. PMID 14597768